CLINICAL TRIAL: NCT02688166
Title: Cardiac Magnetic Resonance Imaging and Biomarker Testing for Evaluating Cardiac Injury Resulting From Radiation Therapy in Cancer: A Pilot Study
Brief Title: Cardiac MRI Biomarker Testing (GCC 1618)
Status: Terminated | Type: Observational
Why Stopped: Unable to meet accrual goal
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00068503
Record Dates: First submitted 2016-02-12; First posted 2016-02-23 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Lung Cancer (Non-Small Cell); Thoracic Cancer; Thymic Cancer; Mesothelioma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Thymus Neoplasms; Mesothelioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer: Breast cancer patients who are undergoing internal mammary lymph node radiation
  Interventions: Other: Complete Cardiac Magnetic Resonance Imaging (MRI)
- Lung Cancer, thymic cancer or mesothelioma: Non-surgical Stage III non-small cell lung cancer patients undergoing mediastinal nodal irradiation with curative intent using concurrent chemotherapy
  Any lung cancer, thymic cancer or mesothelioma patient getting either chemoradiation or radiation alone wherein heart gets radiation exposure
  Interventions: Other: Complete Cardiac Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Complete Cardiac Magnetic Resonance Imaging (MRI) — Complete Cardiac Magnetic Resonance Imaging (MRI) prior to treatment and then at approximately 1 year after completion of radiation therapy

SUMMARY:
This research study can help understand how cardiac changes may occur with radiation therapy to the heart based off measurements obtained through biomarkers and cardiac imaging.

Researchers plan to perform cardiac imaging and biomarkers for any cardiac injury. Cardiac magnetic resonance imaging (CMR) provides the ability to quantitatively measure cardiac function and injury. The cardiac biomarkers that will be tested are effective in the diagnosis, risk-stratification, and monitoring of heart failure.

DETAILED DESCRIPTION:
The goal is to assess the validity of CMR and biomarker examinations before and after radiotherapy for lung cancer, thymic cancer, mesothelioma and breast cancers will demonstrate evidence of cardiac strain and dysfunction proportional to the extent of cardiac exposure during the course of radiation. The investigators intention is to conduct a pilot study of 10 patients receiving moderate doses of radiation exposure to the heart (5 lung cancer patients, , thymic cancer or mesothelioma and 5 breast cancer patients) when treated by our current institutional standards with the idea that this could lead to a grant if early signs of cardiac injury can be measured. These patients' treatment plans would include contours to measure dose received by multiple structures within the heart (coronary vessels and all cardiac chambers) as well as the heart/pericardium itself. The investigators would obtain biomarkers by bloodwork before, during, and after radiotherapy for correlation with clinical outcomes and Cardiac MRIs obtained prior to and 1 year after completion of radiotherapy. Investigators would obtain biomarkers by bloodwork before, during, and after radiotherapy for correlation with clinical outcomes and Cardiac MRs obtained prior to and 1 year after completion of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who are undergoing internal mammary lymph node radiation which is the investigators institutional policy for patients with axillary lymph node involvement
* Clinical AJCC (AJCC, 7th ed.) II, IIIA or IIIB with non-operable disease or those who refuse surgery who are recommended concurrent chemoradiation. Patients who present with N2 or N3 disease and an undetectable NSCLC primary tumor are eligible.
* Any lung cancer, thymic cancer or mesothelioma patient getting either chemoradiation or radiation alone wherein heart gets radiation exposure
* Patients who have received systemic treatment (up to 4 cycles of induction chemotherapy, or up to 6 months of targeted therapy) and are rendered candidate for concurrent chemoradiation are also eligible
* Patients with recurrent disease overlapping or in close proximity to heart getting hypofractionated or conventionally fractionated proton therapy alone.
* Intensity modulated radiotherapy, 3-D conformal radiotherapy, electron radiotherapy, and proton radiotherapy will be permitted.
* Patients who develop local or nodal recurrence after surgery and rendered candidate for definitive concurrent chemoradiation are also eligible.
* The patient must give protocol-specific consent on an IRB approved consent form prior to completion of protocol specific testing/procedures.
* 18 years of age or older.

Exclusion Criteria:

* Pregnant/breast feeding patients or those not willing to undertake contraception if of child-producing potential while on study
* Patients with Stage IV disease
* Patients with contraindications to MRI examination (e.g. gadolinium allergies/reactions, metallic implants, incompatible implanted electronic/cardiac devices, over scanner weight tolerance etc.)
* Patients with hepatorenal syndrome
* Patients with Chronic Kidney Disease defined as eGFR <30 ml/min
* Patients unable to lie supine for 30 minutes for MRI examination
* Patients having undergone prior radiation therapy to the chest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators hypothesize that CMR and biomarker examinations before and after radiotherapy for lung cancer, thymic cancer or mesothelioma and breast cancers will demonstrate evidence of cardiac strain and dysfunction proportional to the extent of cardiac exposure during the course of radiation. Investigators intent to conduct a pilot study of 10 patients receiving moderate doses of radiation exposure to heart (5 lung cancer, thymic cancer, mesothelioma and 5 breast cancer patients) when treated by our current institutional standards with the idea that this could lead to a grant if early signs of cardiac injury can be measured. These patients' treatment plans would include contours to measure dose received by multiple structures within the heart (coronary vessels and all cardiac chambers) as well as the heart/pericardium itself.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Evaluate for evidence of changes in cardiac function measured by cardiac MRI prior to and following external beam radiotherapy who are receiving moderate doses of radiation to the heart. | Baseline and 2 years
Evidence of changes in cardiac function as measured by serum biomarkers following external beam radiotherapy who are receiving moderate doses of radiation to the heart. | Baseline and 2 years

SECONDARY OUTCOMES:
Correlate changes in cardiac function measured by cardiac MRI with radiotherapy dose volume histograms evaluating multiple components of the heart. | Baseline and 2 years
Correlate changes in cardiac function measured by serum biomarkers with radiotherapy dose volume histograms evaluating multiple components of the heart. | Baseline and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Nichols, MD, Principal Investigator — University of Maryland Dept. of Radiation Oncology
Locations (1):
- Ummc Msgccc, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No